CLINICAL TRIAL: NCT00683839
Title: Tobacco Cessation Via Public Health Dental Clinics (PHD2)
Brief Title: Tobacco Cessation Via Public Health Dental Clinics
Acronym: PHD2
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Oregon Research Institute (Other)
Collaborators: Columbia University (Other); University of Mississippi Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 5R01CA107442-3; 5R01CA107442 (NIH)
Record Dates: First submitted 2008-05-16; First posted 2008-05-26 (Estimated); Last update posted 2011-10-26 (Estimated); Status verified 2011-10

CONDITIONS: Smoking
Keywords: Tobacco; Smoking; Smokeless; Cessation; Public health clinic; Dental patients; 5 As; NRT; Tobacco Quit Line; Smokeless tobacco
MeSH Terms: conditions — Smoking; Tobacco Use

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 2 (Experimental): Dental practitioners provide the following intervention:
  5As plus nicotine replacement therapy The 5As consist of: Ask, Advise, Assess, Assist and Arrange.
  Interventions: Behavioral: Brief tobacco counseling
- 1 (No Intervention): Usual Care Control: Patients receive treatment as usual.

INTERVENTIONS:
Behavioral: Brief tobacco counseling — Public health dental professionals provide brief counseling during routine visits based on the Clinical Practice Guidelines 5 As (Ask, Advise, Assess, Assist, Arrange), including offering free Nicotine Replacement Therapy and referral to a Tobacco Quit Line. Pharmacologic: nicotine patch or lozenge maximum 12 week course.
  Arms: 2

SUMMARY:
The study will examine the effectiveness of public health dental practitioners using a brief office based intervention designed to help patients quit smoking or smokeless tobacco use, as compared to usual care.

DETAILED DESCRIPTION:
The prevalence of tobacco use is especially high in lower socioeconomic status (SES) populations in the U.S. Community Health Centers provide comprehensive primary care services, and usually dental services, to large numbers of low-income smokers and smokeless tobacco users. The typical patient has multiple dental visits, which can be used for tobacco cessation advice and counseling by the dental office team. This study builds on a successful pilot study conducted in two public health dental clinics.

This study is a randomized clinical trial in which 14 public health dental clinics in Oregon, Mississippi, and New York City were stratified by state, matched within state by racial/ethnic composition, and then randomly assigned to either the Intervention or Usual Care Control condition. In the Intervention Condition, the dental team provided a brief intervention modeled on the "5A's" advocated by the Clinical Practice Guideline.

ELIGIBILITY:
Inclusion Criteria:

* Patients of participating public health dental clinics
* Tobacco users

Exclusion Criteria:

* Emergency patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2637 (Actual)
Dates: Start 2006-01; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
The primary outcome is prolonged abstinence at 7.5 months following intervention. | 7.5 months

SECONDARY OUTCOMES:
Reduction in tobacco use at 6 weeks and 7.5 months following intervention. | 6 weeks and 7.5 months
Number of quit attempts at 6 weeks and 7.5 months following intervention. | 6 weeks & 7.5 months
Increase in readiness to quit at 6 weeks & 7.5 months following intervention. | 6 weeks & 7.5 months

CONTACTS AND LOCATIONS:
Overall Officials: Judith S. Gordon, Ph.D, Principal Investigator — Oregon Research Institute
Locations (3):
- United States (3):
  - University of Mississippi, Jackson, Mississippi
  - Columbia University, New York, New York
  - Oregon Research Institute, Eugene, Oregon

REFERENCES:
- [Background] Hinds E, Gordon JS, Widdop CJ. Tobacco Cessation in Public Health Dental Clinics: Short-Term Outcomes for Women. Society of Behavioral Medicine's 29th Annual Meeting and Scientific Sessions in San Diego, California, March 26-29th, 2008.
- [Result] Gordon JS, Andrews JA, Albert DA, Crews KM, Payne TJ, Severson HH. Tobacco cessation via public dental clinics: results of a randomized trial. Am J Public Health. 2010 Jul;100(7):1307-12. doi: 10.2105/AJPH.2009.181214. Epub 2010 May 13. PMID 20466951
- [Derived] Theodoulou A, Fanshawe TR, Leavens E, Theodoulou E, Wu AD, Heath L, Stewart C, Nollen N, Ahluwalia JS, Butler AR, Hajizadeh A, Thomas J, Lindson N, Hartmann-Boyce J. Differences in the effectiveness of individual-level smoking cessation interventions by socioeconomic status. Cochrane Database Syst Rev. 2025 Jan 27;1(1):CD015120. doi: 10.1002/14651858.CD015120.pub2. PMID 39868569
- [Derived] Holliday R, Hong B, McColl E, Livingstone-Banks J, Preshaw PM. Interventions for tobacco cessation delivered by dental professionals. Cochrane Database Syst Rev. 2021 Feb 19;2(2):CD005084. doi: 10.1002/14651858.CD005084.pub4. PMID 33605440